CLINICAL TRIAL: NCT07291479
Title: Development of Upper Extremity Behavioral Assessment Methods for Reach-and-grasp and Physical Rehabilitation.
Brief Title: Behavioral Assessment Method Index
Acronym: BAM
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Professor, Ohio State University
Other Study IDs: 2021H0419
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-01

CONDITIONS: Infant Development; Perinatal Stroke; Hemiparesis; Cerebral Palsy
MeSH Terms: conditions — Paresis; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Typically developing infants
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Prospective sample is typically developing. No intervention.

SUMMARY:
The overall goal of this study is to develop and improve assessment methods for children with and without perinatal arterial ischemic stroke (PAS)/hemiparetic cerebral palsy (HCP). The focus is on behaviors of the arms and hands and includes other domains of child development like fine motor, gross motor, language, cognition, and social-emotional skills. This study involves 1) the use of data, including video recordings, from "I-ACQUIRE - Perinatal Arterial Stroke: A Multi-site RCT of Intensive Infant Rehabilitation" (NCT03910075) and 2) a prospective longitudinal observational data collection with a typically developing cohort using a comprehensive assessment battery (play, fine motor, gross motor, language, cognition, and social emotional skills). The current study is called the BAM Index. No intervention or treatment is provided as part of the BAM Index. The I-ACQUIRE study is an RCT that includes an intervention. The BAM index study is a use of data from the I-ACQUIRE cohorts and a prospective observational study of a typically developing cohort (children without stroke or cerebral palsy) over time. The results of this work will develop, test, refine, and validate a new methodology based on reach-and-grasp and other behaviors related to child development that will have profound and lasting impact on assessment and selection of treatment strategies for pediatric physical rehabilitation of children. The use and reuse of video technology is also well-suited to remote or virtual assessment. This proposal will add to our current knowledge by 1) yielding a psychometrically robust and alternative approach to measuring upper extremity function in children with stroke and/or hemiparetic cerebral palsy and 2) defining specific parameters about how to promote closer-to-normal upper extremity function in children with motor disability.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 36 months old at baseline
* Full Term Birth (37 to 41 weeks gestation)
* Healthy development (meeting age-appropriate milestones)

Exclusion Criteria:

* Diagnosed or suspected impairments (auditory, visual, cognitive or motor)

Ages: 4 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy, typically developing children, born at full-term.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Behavioral Assessment Methods (BAM) | From enrollment to the last assessment (7 months).
  Calculated based on reach- and grasp parameters with a variety of object explorations.

SECONDARY OUTCOMES:
How the BAM index is related to fine motor, gross motor, cognition, and language skills across development for typical and atypical infants. | From enrollment to the last assessment (7 months).
  Clinician and parent collected standardized measures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No